CLINICAL TRIAL: NCT07037667
Title: Effect of Pilates Exercises in Management of Premenstrual Anxiety
Brief Title: New Management of PMS Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Summer Kamal Abbas Mabrouk, Master's degree student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004060
Record Dates: First submitted 2025-06-10; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-10

CONDITIONS: Premenstrual Anxiety
Keywords: Premenstrual; Anxiety; Pilates exercises
MeSH Terms: conditions — Anxiety Disorders | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): This group will do Pilates exercises as single leg lift 10 rep and one leg circle 5 times in each direction for 15 minutes 2 times per week for 12 weeks and receives dietary recommendations as healthy snacks that are rich in magnesium and vitamin B-6.
  Interventions: Other: Pilates exercises; Other: Dietary recommendations
- Control group (Placebo Comparator): This group will receive dietary recommendations as healthy snacks that are rich in magnesium and vitamin B-6.
  Interventions: Other: Dietary recommendations

INTERVENTIONS:
Other: Pilates exercises — Single leg lifts:The participant is in supine lying position with knees bent and feet parallel and hip-width apart. Head, neck and shoulders totally relaxed and arm extended and relaxed beside the body. Then the participant is asked to inhale first without moving her leg then exhale while bringing one leg up towards chest , drawing her pelvic floor and abdominals up and in like gently tightening a belt and maintaining 90 degrees angle at the knee and then put her leg down while inhaling. One leg circle:The participant is in supine lying position with one leg raised towards the ceiling and the other leg on the floor and both knees slightly bent.Then the participant is asked to inhale first without moving her leg and to make sure to use the abdominal muscles to try to maintain a neutral pelvis while doing the exercise then makes a small circle while exhaling and inhale when she completes the circle and reaches the starting position.
  Arms: Experimental group
Other: Dietary recommendations — Dietary recommendations as healthy snacks that are rich in magnesium and vitamin B-6.

SUMMARY:
The goal of this clinical trial is to determine the effect of Pilates exercises in management of premenstrual anxiety in adult virgin females.The main question it aims to answer is :

Do Pilates exercises have an effect on premenstrual anxiety? Researcher will compare the effect of Pilates exercises to dietary recommendations as healthy snacks rich in magnesium and vitamin B-6 to see if Pilates exercises have an effect on premenstrual anxiety.

Participants will :

Do Pilates exercises two times per week for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All participants are virgins.
* All of them suffering from moderate and severe premenstrual anxiety.
* Their BMI is less than 30 km/m2
* The regularity of their menstrual cycle is 28-35 days.

Exclusion Criteria:

* Smoking.
* Taking any medications for anxiety.
* Irregular menstruation.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2024-05-22 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Change in premenstrual anxiety | 12 weeks following end of treatment
  State-Trait- Anxiety Inventory for adults (STAI-AD)

CONTACTS AND LOCATIONS:
Locations (1):
- Elbeheira governorate, Damanhūr, Egypt

IPD SHARING:
Plan to Share IPD: No